CLINICAL TRIAL: NCT05151471
Title: A Phase 3b, Multicenter, Randomized, Double-blind Extension Study to Evaluate the Continued Efficacy and Safety of Oral Edaravone Administered for an Additional Period of up to 48 Weeks Following Study MT-1186-A02 in Subjects With Amyotrophic Lateral Sclerosis (ALS)
Brief Title: Efficacy and Safety Extension Study of Oral Edaravone Administered in Subjects With ALS
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Futility Analysis of parent study MT-1186-A02 was met.
Sponsor: Tanabe Pharma America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MT-1186-A04; jRCT2071210117 (Registry Identifier: Japan Registry of Clinical Trials (jRCT)); 2021-003900-42 (EudraCT Number)
Record Dates: First submitted 2021-11-28; First posted 2021-12-09 (Actual); Results first posted 2025-03-27 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: ALS
MeSH Terms: interventions — Edaravone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- MT-1186 - Group 1 (Experimental): Oral edaravone administered once daily for up to 48 weeks or until the drug is commercially available in that country.
  Interventions: Drug: MT-1186
- MT-1186 - Group 2 (Experimental): Oral edaravone administered for 10 days followed by 18-day placebo (regimen denoted as on/off) for up to 48 weeks or until the drug is commercially available in that country.
  Interventions: Drug: MT-1186; Drug: Placebo

INTERVENTIONS:
Drug: MT-1186 — Oral edaravone
  Other Names: Oral edaravone
Drug: Placebo — Oral
  Other Names: Oral
  Arms: MT-1186 - Group 2

SUMMARY:
To evaluate and compare the efficacy of two dosing regimens of oral edaravone in subjects with amyotrophic lateral sclerosis (ALS), based on the time from the randomization date in Study MT-1186-A02 to at least a 12-point decrease in Revised ALS Functional Rating Score (ALSFRS-R) or death, whichever happens first, over the course of the study or until oral edaravone is commercially available in that country

ELIGIBILITY:
Inclusion Criteria:

1. Subjects or their legally authorized representative must provide a signed and dated informed consent form to participate in the study.
2. Subjects must be able (in the judgment of the Investigator) to understand the nature of the study and all risks involved with participation in the study.
3. Subjects must be willing to cooperate and comply with all protocol restrictions and requirements.
4. Subjects must have successfully completed all Study MT-1186-A02 visits and have been compliant with study drug.

Exclusion Criteria:

1. Subjects of childbearing potential unwilling to use an acceptable method of contraception from the Day 1/screening visit until 3 months after the last dose of study medication. Subjects who are sexually active who do not agree to use contraception during the study period.
2. Subjects who are female, of childbearing potential, and pregnant (a positive pregnancy test) or lactating at the Day 1/screening visit.
3. Subjects who have a significant risk of suicide. Subjects with any suicidal behavior or suicidal ideation of type 4 (active suicidal ideation with some intent to act, without a specific plan) or type 5 (active suicidal ideation with specific plan and intent) based on the Columbia-Suicide Severity Rating Scale (C-SSRS) at Week 48 of Study MT-1186-A02.
4. Subjects who are not eligible to continue in the study, as judged by the Investigator in conjunction with the MTDA medical monitor.
5. Subjects who are unable to take their medications orally or through a PEG/RIG tube.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 202 (Actual)
Dates: Start 2022-01-11 (Actual); Primary Completion 2023-09-29 (Actual); Study Completion 2023-09-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Head of Medical Science, Study Director — Tanabe Pharma America, Inc.
Locations (37):
- United States (10):
  - Woodland Research Northwest, LLC, Rogers, Arkansas
  - UF Health Cancer Center/Clinical Trials Office, Gainesville, Florida
  - Emory University - School of Medicine, Atlanta, Georgia
  - Northwestern University Feinberg School of Medicine, Chicago, Illinois
  - Johns Hopkins University, Baltimore, Maryland
  - Neurology Associates, P.C - Lincoln, Lincoln, Nebraska
  - University Of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Nerve And Muscle Center Of Texas, Houston, Texas
  - University of Washington Medical Center, Seattle, Washington
  - West Virginia University School of Medicine (WVUSoM) - Movement Disorder Clinic, Morgantown, West Virginia
- Canada (4):
  - University of Alberta - Walter C Mackenzie Health Sciences Centre (WCM), Edmonton, Alberta
  - Health Science Center Mcmaster University, Hamilton, Ontario
  - London Health Sciences Centre - University Hospital, London, Ontario
  - CHU de Quebec-Hopital-Enfant-Jesus, Québec, Quebec
- Universitaetsklinikum Wuerzburg, Würzburg, Germany
- Japan (20):
  - National Hospital Organization Higashinagoya National Hospital, Nagoya, Aichi-ken
  - Nagoya University Hospital, Nagoya, Aichi-ken
  - National Hospital Organization Chibahigashi National Hospital, Chiba, Chiba
  - Murakami Karindoh Hospital, Fukuoka, Fukuoka
  - Fukushima Medical University Hospital, Fukushima, Fukushima
  - Hiroshima University Hospital, Hiroshima, Hiroshima
  - National Hospital Organization Iou National Hospital, Kanazawa, Ishikawa-ken
  - Kagawa University Hospital, Kita-gun, Kagawa-ken
  - Yokohama City University Hospital, Yokohama, Kanagawa
  - National Hospital Organization Kumamoto Saishun Medical Center, Kōshi, Kumamoto
  - National Hospital Organization Utano National Hospital, Kyoto, Kyoto
  - Tohoku University Hospital, Sendai, Miyagi
  - Niigata University Medical & Dental Hospital, Niigata, Niigata
  - Kansai Electric Power Hospital, Osaka, Osaka
  - National Hospital Organization Osaka Toneyama Medical Center, Toyonaka, Osaka
  - National Hospital Organization Shizuoka Institute of Epilepsy and Neurological Disorders, Shizuoka, Shizuoka
  - Tokyo Metropolitan Neurological Hospital, Fuchū, Tokyo
  - Teikyo University Hospital, Itabashi-ku, Tokyo
  - Toho University Omori Medical Center, Ōta-ku, Tokyo
  - Saitama Neuropsychiatric Institute, Saitama
- Hanyang University Medical Center, Wangsimni-ro, Seongdong-gu, South Korea
- Chefarzt Muskelzentrum/ALS Clinic Kantonsspital St.Gallen Muskelzentrum/ALS Clinic, Sankt Gallen, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- Edaravone 105 mg (Once Daily): Oral edaravone administered once daily for up to 48 weeks or until the drug is commercially available in that country.
  MT-1186: Oral edaravone
- Edaravone 105 mg (on/Off): Oral edaravone administered for 10 days followed by 18-day placebo (regimen denoted as on/off) for up to 48 weeks or until the drug is commercially available in that country.
  MT-1186: Oral edaravone
  Placebo: Oral
Period: Overall Study
Arm/Group | Edaravone 105 mg (Once Daily) | Edaravone 105 mg (on/Off)
Started | 104 | 98
Completed | 24 | 24
Not Completed | 80 | 74
Not completed — Adverse Event | 21 | 16
Not completed — Death | 1 | 0
Not completed — Lost to Follow-up | 0 | 1
Not completed — Withdrawal by Subject | 7 | 9
Not completed — Study terminated by sponsor | 49 | 47
Not completed — Other | 2 | 1

BASELINE CHARACTERISTICS:
Population: The data collected before the first study drug dose administration date in Study MT-1186-A02 will be used as the baseline for statistical analysis in Study MT-1186-A04.
Groups:
- Total: Total of all reporting groups
Arm/Group | Edaravone 105 mg (Once Daily) | Edaravone 105 mg (on/Off) | Total
Number analyzed (Participants) | 192 | 192 | 384
Age, Customized [Count of Participants; unit: Participants]
  Adults (18-64 years) | 134 | 122 | 256
  From 65-84 years | 58 | 70 | 128
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 69 | 70 | 139
  Male | 123 | 122 | 245
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 115 | 109 | 224
  Black or African American | 3 | 2 | 5
  Asian - Japanese | 63 | 64 | 127
  Asian - Not Japanese | 8 | 13 | 21
  American Indian or Alaska Native | 0 | 1 | 1
  Native Hawaiian or Pacific Islander | 0 | 1 | 1
  Not Reported | 0 | 1 | 1
  Other | 3 | 1 | 4

OUTCOME MEASURES:

1. Primary Outcome: Time From the Randomization Date in Study MT-1186-A02 to at Least a 12-point Decrease in ALSFRS-R or Death, Whichever Happens First.
Description: The ASLFRS-R is Amyotrophic Lateral Sclerosis Functional Rating Scale-Revised. The ALSFRS-R measures 12 aspects of physical function, ranging from one's ability to swallow and use utensils to climbing stairs and breathing. Each function is scored from 4 (normal) to 0 (no ability), with a maximum total score of 48 and a minimum total score of 0.
Time Frame: Up to 96 weeks
Population: The outcome measure time frame is from the randomization date in Study MT- 1186-A02 to at least a 12-point decrease in ALSFRS-R or death, whichever happened first.
Measure: Mean (80% Confidence Interval); unit: Month
Arm/Group | Edaravone 105 mg (Once Daily) | Edaravone 105 mg (on/Off)
Number analyzed (Participants) | 192 | 192
Month | 13.9 [13.4 to 16.59] | 15.05 [13.8 to 16.62]
Statistical Analysis 1: Comparison: Edaravone 105 mg (Once Daily) vs Edaravone 105 mg (on/Off); Test type: Superiority; p = 0.78, Log Rank

2. Secondary Outcome: The Combined Assessment of Function and Survival (CAFS) Score at All Visits From Baseline in Study MT-1186-A02 to the End of Study MT-1186-A04
Description: CAFS analysis ranks clinical outcomes on the basis of survival time and change in the ALS Functional Rating Scale-Revised (ALSFRS-R) score. A subject's score will be calculated by comparing each subject to every other subject within each treatment group in the study, resulting in a score of +1 if the outcome was better than the subject being compared, -1 if worse, and 0 if the same. The subject's score will then be calculated by summing up their comparison to all of the other subjects within each treatment group in the study as CAFS score. Patients' summary scores are ranked; a higher score indicates a better performance. The score range is from 1 to N, where N is the total sample size.
  Since CAFS were calculated using the imputed ALSFRS-R scores with multiple imputation method, and the maximum varies for each simulation, 383 is the maximum possible value of full range for measure of dispersion.
Time Frame: Baseline, Week 72 and Week 96
Population: One subject randomized to the On/Off treatment group was excluded from this analysis because the subject did not receive any study treatment.
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Edaravone 105 mg (Once Daily) | Edaravone 105 mg (on/Off)
Number analyzed (Participants) | 192 | 191
units on a scale
  Week 72 | 193.6 [4 to 383] | 189.1 [1 to 383]
  Week 96 | 200.8 [4 to 383] | 181.6 [1 to 383]
Statistical Analysis 1: Comparison: Edaravone 105 mg (Once Daily) vs Edaravone 105 mg (on/Off); Week 72; Test type: Superiority; p = 0.704, ANCOVA
Statistical Analysis 2: Comparison: Edaravone 105 mg (Once Daily) vs Edaravone 105 mg (on/Off); Week 96; Test type: Superiority; p = 0.131, ANCOVA

3. Secondary Outcome: Change in the Amyotrophic Lateral Sclerosis Assessment Questionnaire 40 Score at All Visits From Baseline in Study MT-1186-A02 to the End of Study MT-1186-A04
Description: The ALSAQ-40 is a questionnaire that consists of 40 questions/items with 5 discrete scales: physical mobility, activities of daily living and independence, eating and drinking, communication, emotional reactions, ranging from 0 (best health as assessed by the scale) to 100 (worse health as assessed by the measure).
Time Frame: Baseline, Week 72 and Week 96
Population: Those patients reached to Week 72 and Week 96, and conducted ALSAQ-40 assessment.
Measure: Least Squares Mean (Standard Error); unit: Point
Arm/Group | Edaravone 105 mg (Once Daily) | Edaravone 105 mg (on/Off)
Number analyzed (Participants) | 192 | 191
Point
  Week 72: number analyzed (Participants) | 67 | 72
  Week 72 | 45.71 (3.14) | 45.46 (3.11)
  Week 96: number analyzed (Participants) | 31 | 27
  Week 96 | 54.83 (4.05) | 57.91 (4.13)
Statistical Analysis 1: Comparison: Edaravone 105 mg (Once Daily) vs Edaravone 105 mg (on/Off); Week 72; Test type: Superiority; p = 0.954, Mixed Model for Repeated Measures (MMRM)
Statistical Analysis 2: Comparison: Edaravone 105 mg (Once Daily) vs Edaravone 105 mg (on/Off); Week 96; Test type: Superiority; p = 0.591, Mixed Model for Repeated Measures (MMRM)

4. Secondary Outcome: Change in ALSFRS-R Score at All Visits From Baseline in Study MT-1186-A02 to the End of Study MT-1186-A04
Description: The ALSFRS-R is rating scale (ratings 0 = can't do, to 4 = normal ability) used to determine participants' assessment of their capability and independence in 12 functional activities.
Time Frame: Baseline, Week 72, Week 84 and Week 96
Population: Those patients reached to Week 72, Week 84 and Week 96, and conducted ALSFRS-R assessment.
Measure: Least Squares Mean (Standard Error); unit: Point
Arm/Group | Edaravone 105 mg (Once Daily) | Edaravone 105 mg (on/Off)
Number analyzed (Participants) | 192 | 191
Point
  Week 72: number analyzed (Participants) | 67 | 74
  Week 72 | -15.02 (0.95) | -15.90 (0.95)
  Week 84: number analyzed (Participants) | 46 | 49
  Week 84 | -16.79 (1.11) | -18.27 (1.10)
  Week 96: number analyzed (Participants) | 31 | 29
  Week 96 | -18.21 (1.31) | -20.95 (1.32)
Statistical Analysis 1: Comparison: Edaravone 105 mg (Once Daily) vs Edaravone 105 mg (on/Off); Week 72; Test type: Superiority; p = 0.513, Mixed Model for Repeated Measures (MMRM)
Statistical Analysis 2: Comparison: Edaravone 105 mg (Once Daily) vs Edaravone 105 mg (on/Off); Week 84; Test type: Superiority; p = 0.344, Mixed Model for Repeated Measures (MMRM)
Statistical Analysis 3: Comparison: Edaravone 105 mg (Once Daily) vs Edaravone 105 mg (on/Off); Week 96; Test type: Superiority; p = 0.142, Mixed Model for Repeated Measures (MMRM)

5. Secondary Outcome: Time From the Randomization Date in Study MT-1186-A02 to Death, Tracheostomy, or Permanent Assisted Mechanical Ventilation (≥23 Hours/Day)
Time Frame: Up to 96 weeks
Population: The outcome measure time frame is from Baseline in Study MT-1186-A02 to the End of Study MT-1186-A04.
Measure: Median (95% Confidence Interval); unit: Month
Arm/Group | Edaravone 105 mg (Once Daily) | Edaravone 105 mg (on/Off)
Number analyzed (Participants) | 192 | 192
Month | NA [19.36 to 21.02] — The median survival for the time to death could not be calculated due to the low number of events (only 33 and 32 events of death, tracheostomy, or PAMV in the Once Daily and On/Off groups, respectively), resulting in 159 and 160 censored observations in respective group (i.e., NA means NE (Not estimable)). | NA [19.43 to 21.13] — The median survival for the time to death could not be calculated due to the low number of events (only 33 and 32 events of death, tracheostomy, or PAMV in the Once Daily and On/Off groups, respectively), resulting in 159 and 160 censored observations in respective group (i.e., NA means NE (Not estimable)).

6. Secondary Outcome: Time From the Randomization Date in Study MT-1186-A02 to Death or Permanent Assisted Mechanical Ventilation (>23 Hours/Day)
Time Frame: Up to 96 weeks
Population: The outcome measure time frame is from Baseline in Study MT-1186-A02 to the End of Study MT-1186-A04.
Measure: Median (95% Confidence Interval); unit: Month
Arm/Group | Edaravone 105 mg (Once Daily) | Edaravone 105 mg (on/Off)
Number analyzed (Participants) | 192 | 192
Month | NA [NA to NA] — The median survival for the time to death could not be calculated due to the low number of events (only 30 and 31 events of death or PAMV in the Once Daily and On/Off groups, respectively), resulting in 162 and 161 censored observations in respective group (i.e., NA of Median means NE (Not estimable)). | NA [NA to NA] — The median survival for the time to death could not be calculated due to the low number of events (only 30 and 31 events of death or PAMV in the Once Daily and On/Off groups, respectively), resulting in 162 and 161 censored observations in respective group (i.e., NA of Median means NE (Not estimable)).

7. Secondary Outcome: Time From the Randomization Date in Study MT-1186-A02 to Death
Time Frame: Up to 96 weeks
Population: The outcome measure time frame is from Baseline in Study MT-1186-A02 to the End of Study MT-1186-A04.
Measure: Median (95% Confidence Interval); unit: Month
Arm/Group | Edaravone 105 mg (Once Daily) | Edaravone 105 mg (on/Off)
Number analyzed (Participants) | 192 | 192
Month | NA [NA to NA] — The median survival for the time to death could not be calculated due to the low number of events (only 24 and 28 events of death in the Once Daily and On/Off groups, respectively), resulting in 168 and 164 censored observations in respective group (i.e., NA of Median means NE (Not estimable)). | NA [NA to NA] — The median survival for the time to death could not be calculated due to the low number of events (only 24 and 28 events of death in the Once Daily and On/Off groups, respectively), resulting in 168 and 164 censored observations in respective group (i.e., NA of Median means NE (Not estimable)).

ADVERSE EVENTS:
Time Frame: Up to 50 weeks
Description: All AEs and SAEs that occur from the time written ICF was obtained until the end of the Safety Follow-up Period or the withdrawal of the subject from the study. The All-Causes Mortality time frame is from Day1 to the End of study MT-1186-A04. On the other hand, time frame of Outcome Measure 7 is from Day1 in MT-1186-A02 to the End of study MT-1186-A04. Therefore, the number of participants of death (i.e., "15" and "12") is inconsistent with information in the NA Explanation in Outcome Measure 7.
Arm/Group | Edaravone 105 mg (Once Daily) | Edaravone 105 mg (on/Off)
All-Cause Mortality (participants affected / at risk) | 15/104 | 12/98
Serious Adverse Events (participants affected / at risk) | 33/104 | 27/98
Other Adverse Events (participants affected / at risk) | 24/104 | 25/98
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Edaravone 105 mg (Once Daily) (N=104) | Edaravone 105 mg (on/Off) (N=98)
Cardiac arrest (Cardiac disorders) | 0 | 1
Cardio-respiratory arrest (Cardiac disorders) | 1 | 0
Dysphagia (Gastrointestinal disorders) | 14 | 5
Nausea (Gastrointestinal disorders) | 1 | 0
COVID-19 (Infections and infestations) | 2 | 1
COVID-19 pneumonia (Infections and infestations) | 1 | 0
Catheter site infection (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 2 | 1
Respiratory tract infection viral (Infections and infestations) | 1 | 0
Urosepsis (Infections and infestations) | 1 | 0
Clavicle fracture (Injury, poisoning and procedural complications) | 1 | 0
Extradural haematoma (Injury, poisoning and procedural complications) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 2
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 1
Thermal burn (Injury, poisoning and procedural complications) | 1 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Amyotrophic lateral sclerosis (Nervous system disorders) | 4 | 1
Device dislocation (Product Issues) | 0 | 1
Device malfunction (Product Issues) | 1 | 0
Psychiatric symptom (Psychiatric disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 1
Oliguria (Renal and urinary disorders) | 1 | 0
Urethral stenosis (Renal and urinary disorders) | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Asphyxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Orthopnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 10 | 10
Sputum retention (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Gastrostomy (Surgical and medical procedures) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Edaravone 105 mg (Once Daily) (N=104) | Edaravone 105 mg (on/Off) (N=98)
Constipation (General disorders) | 7 | 6
Diarrhoea (General disorders) | 4 | 5
COVID-19 (Infections and infestations) | 6 | 1
Fall (Injury, poisoning and procedural complications) | 8 | 13
Insomnia (Psychiatric disorders) | 5 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2022-07-29): https://cdn.clinicaltrials.gov/large-docs/71/NCT05151471/Prot_000.pdf
  • Statistical Analysis Plan (2024-01-10): https://cdn.clinicaltrials.gov/large-docs/71/NCT05151471/SAP_001.pdf